CLINICAL TRIAL: NCT02646553
Title: Saliva Cortisol Measurement as a Screening Test for Suspicious Cushings Syndrome in Children.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2012/842
Record Dates: First submitted 2016-01-04; First posted 2016-01-05 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Cushings Syndrome
MeSH Terms: conditions — ACTH Syndrome, Ectopic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — the investigators collect saliva and urine from the patients, for analysis of the hormone cortisol.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Children refered to the obesity clinic.: All children refered to the obesity clinic for examination and optionally treatment are invited.
  Interventions: Other: Children refered to the obesity clinic

INTERVENTIONS:
Other: Children refered to the obesity clinic — Compere if urine cortisol is as good as saliva cortisol as a screening for hypercortisolism in children.

SUMMARY:
Cortisol overproduction ( Cushings syndrome) is a condition where the patient have a special fat distribution, with accumulation of fat around the abdomen and in the neck, with thinner limbs and weak musculature. The condition can be difficult to separate from adipositas in general. Screening for hypercortisolism in adults has been easier the last years, because we can measure free cortisol in saliva samples at late night. In children we still dont have reference ranges for saliva cortisol in children, so the screening is still troublesome, based on Collection of 24-hour urine.The meaning of this study is to establish reference ranges for saliva cortisol, and evaluate in a cohort with adipose children if screening with saliva cortisol is sensitive and specific enough to be the New screening test for hypercortisolism in children too.

DETAILED DESCRIPTION:
the investigators have collected saliva samples morning and late evening for cortisol measurements in a total of 330 children ( 660 samples) in the age from 4 to 16 years ols. This samples are going to be used to define a reference range for saliva cortisol in children.

The investigators are then collecting 24 hour urine and saliva samples ( morning and late evening) from children at the obesity clinic Haukeland University hospital for verification of the reference range , and to estimate if the test is good enough to identify the patients that have Cushings syndrome.

Since the diagnose is very seldom in children, we will get help from a 3. line referral center in London to include patients with true Cushings syndrome.

ELIGIBILITY:
Inclusion Criteria:Children aged 4-16 years. Healthy population from selected kindergarten and Schools, and patients refered to the obesity clinic Haukeland University Hospital, for examination and optionally treatment.

-

Exclusion Criteria:Use of any kind of steroids ( oral, liniments, inhalations etc)

-

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The reference are made from healthy children included from kindergarden and Schools in the Bergen area. The age range from 4 to 16 years ols. The patient population is children refered to the obestity clinic at Haukeland University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2012-05; Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Number of patients with positive saliva cortisol measurement, not having Cushings syndrome. | 2 years
  Number of patients
Number of patients With negative saliva cortisol measurement , having Cushings syndrome. | 2 years
  Number of patients

CONTACTS AND LOCATIONS:
Overall Officials: Grethe Åstrøm Ueland, MD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Norway